CLINICAL TRIAL: NCT01296360
Title: Long-Term Immunity and Safety With or Without a Booster Dose Following Primary Vaccination With the Japanese Encephalitis Vaccine IC51 (IXIARO®) in a Pediatric Population in a JEV-Endemic Country. Open-Label, Randomized, Phase 3 Study
Brief Title: Open-label, Randomized Study in a Pediatric Population in a JEV (Japanese Encephalitis Virus)-Endemic Country
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IC51-325
Record Dates: First submitted 2010-12-28; First posted 2011-02-15 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Japanese Encephalitis
Keywords: immune response; IC51-325; Japanese Encephalitis; Intercell AG
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- >14 months to <2 years (Active Comparator): IXIARO 0.25 ml i.m. (milliliter, intramuscular)
  Interventions: Biological: IXIARO
- >3 years - <18 years (Active Comparator): IXIARO 0.5 ml i.m (milliliter, intramuscular)
  Interventions: Biological: IXIARO

INTERVENTIONS:
Biological: IXIARO — 0.25 ml i.m. (milliliter, intramuscular)
  Arms: >14 months to <2 years
Biological: IXIARO — 0.5 ml i.m. (milliliter, intramuscular)
  Arms: >3 years - <18 years

SUMMARY:
This is a randomized, open-label Phase 3 study including children aged >9 months to <17 years and 7 months who have been vaccinated with IXIARO in study IC51-323.

DETAILED DESCRIPTION:
This is a randomized, open-label Phase 3 study including children aged >9 months to <17 years and 7 months who have been vaccinated with IXIARO in the previous study IC51-323.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents who have completed study IC51-323 and received both IXIARO vaccinations according to protocol.
* Children who have received the dose confirmed for their age group.
* Male or female healthy children and adolescents aged ≥9 months to <17 years and 7 months at the time of enrolment into this study.
* Written informed consent by the subject's legal representative(s), according to local requirements, and written informed assent of the subject, if applicable.
* Female subjects: either no childbearing potential or negative pregnancy test (pregnancy test to be performed in female subjects after onset of menarche) at Visits 1, 2 and 2a as stipulated by the protocol. For females after menarche willingness to practice a reliable method of contraception

Exclusion Criteria:

* Vaccination against JE virus (JEV) (except within study IC51-323 and IC51 325), Yellow fever, West Nile virus and Dengue fever at any time prior to or planned during the study.
* History of or clinical manifestation of any Flavivirus disease during IC51-323 or IC51 325.
* Participation in another study with an investigational drug during IC51 323 or IC51 325.
* Planned active or passive immunization within 2 weeks before and 1 week after the IXIARO booster.
* History of or development of any immunodeficiency including post-organ-transplantation after inclusion into IC51-323 or IC51 325.
* History of or development of an autoimmune disease during study IC51-323 or IC51 325.

  * Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying medications started during IC51-323 or IC51 325. (For corticosteroids, this would mean prednisone or equivalent at >0.05 mg/kg/day; topical and inhaled steroids are allowed).
* Acute febrile infection at Visit 2 (only for the Booster Group).
* Pregnancy (positive pregnancy test at Visit 1 and Visit 2), lactation or unreliable contraception in female subjects after onset of menarche.
* Hypersensitivity reactions to IXIARO or adverse events in study IC51-323 requiring withdrawal from further vaccination or anaphylaxis or severe cases of atopy requiring emergency treatment or hospital admission during IC51-323 or IC51 325.
* History of urticaria after hymenoptera envenomation, drugs, physical or other provocations or of idiopathic cause during IC51-323 or IC51 325.
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) (measurement of Hepatitis B surface antigen [HBsAg] titers) or hepatitis C virus (HCV).
* Illicit drug use and/or current drug or alcohol addiction.
* Inability or unwillingness by the legal representative(s) and/or the subject (where applicable) to provide informed consent/assent and to abide by the requirements of the study.
* Persons who have been committed to an institution (by a court or by an authority).

Ages: 9 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Kadlecek, Mag., Study Chair — Valneva Austria GmbH
Locations (3):
- Philippines (3):
  - Research Institute for Tropical Medicine - Clinical Research Division, City of Muntinlupa, Alabang
  - Research Institute for Tropical Medicine, City of Muntinlupa, Alabang
  - UP-Philippine General Hospital, Manila, Manila

RESULTS

PARTICIPANT FLOW:
Groups:
- Booster Group: IC51 booster vaccination ~12 months after primary immunization in study IC51-323
- Non-Booster Group: No treatment in study IC51-325
Period: Overall Study
Arm/Group | Booster Group | Non-Booster Group
Started | 150 | 150
Visit 2 (Month 12) | 148 (booster was administered) | 149
Visit 2a (Month 13) | 148 (visit in Booster Group only: ~13 months after immunization in IC51-323 (i.e., 1 month post booster)) | 0
Completed | 144 | 142
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Population: Safety Population: subjects who entered into the study and were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Booster Group | Non-Booster Group | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.23 (5.084) | 5.36 (5.135) | 5.30 (5.101)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 79 | 151
  Male | 78 | 71 | 149

OUTCOME MEASURES:

1. Primary Outcome: SCRs (Seroconversion Rate) as Defined by Percentage of Subjects With Plaque Reduction Neutralization Test Titers of>1:10 at 1 Month After the Booster Dose
Time Frame: 1 month post booster
Population: Intent-to-treat Population: primary analysis population for the immunogenicity analyses; defined as all subjects randomized
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- >14 Months to <2 Years: booster vaccination: IXIARO 0.25 ml i.m. (milliliter, intramuscular)
- >3 Years - <18 Years: booster vaccination: IXIARO 0.5 ml i.m (milliliter, intramuscular)
Arm/Group | >14 Months to <2 Years | >3 Years - <18 Years
Number analyzed (Participants) | 81 | 67
percentage of subjects | 100 [95.5 to 100] | 100 [94.6 to 100]

2. Secondary Outcome: Rate of Subjects Achieving a >4-fold Increase in JEV (Japanese Encephalitis Virus) Neutralizing Antibody Titers at 1 Month After the Booster Dose
Time Frame: 1 month
Reporting Status: Not Posted

3. Secondary Outcome: GMTs (Geometric Mean Titre) for JEV Neutralizing Antibodies Measured Using a Validated PRNT (Plaque Reduction Neutralization Test) at 1 Month After the Booster Dose
Time Frame: 1 month
Reporting Status: Not Posted

4. Secondary Outcome: GMTs and Rate of Subjects With a PRNT Titer of >1:10 at Months 12, 24 and 36 After First IXIARO Vaccination in IC51-323 With and Without Booster Vaccination
Time Frame: 36 months
Reporting Status: Not Posted

5. Secondary Outcome: Rate of Subjects With SAEs (Serious Adverse Events) Following Immunization and Medically Attended AEs (Adverse Events) up to Months 12, 24 and 36 After the First IXIARO Vaccination in IC51 323 With and Without Booster Vaccination. Severity, Duration and
Time Frame: 36 months
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Subjects With Unsolicited AEs (Adverse Events) up to Months 12, 24 and 36 After the First IXIARO Vaccination in IC51 323 With and Without Booster Vaccination. Severity, Duration and Relationship to Vaccinations.
Time Frame: 36 months
Reporting Status: Not Posted

7. Secondary Outcome: Rate of Subjects With SAEs and Medically Attended AEs Within 1 Month Following the Booster Dose. Severity, Duration and Relationship to Vaccinations.
Time Frame: 1 month
Reporting Status: Not Posted

8. Secondary Outcome: Rate of Subjects With Unsolicited AEs Within 1 Month Following the Booster Dose. Severity, Duration and Relationship to Vaccinations.
Time Frame: 1 month
Reporting Status: Not Posted

9. Secondary Outcome: Rate of Subjects With Solicited AEs for up to 7 Days Following the Booster Dose. Severity and Duration.
Time Frame: 7 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Booster Group | Non-Booster Group
Serious Adverse Events (participants affected / at risk) | 7/150 | 3/150
Other Adverse Events (participants affected / at risk) | 99/150 | 100/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Booster Group (N=150) | Non-Booster Group (N=150)
Abscess (Infections and infestations) | 1 | 0
Amoebic dysentery (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Paralysis (Nervous system disorders) | 0 | 1
Finger amputation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Booster Group (N=150) | Non-Booster Group (N=150)
Upper respiratory tract infection (Infections and infestations) | 37 | 34
Rhinitis (Infections and infestations) | 17 | 16
Nasopharyngitis (Infections and infestations) | 16 | 15
Varicella (Infections and infestations) | 9 | 14
Gastroenteritis (Infections and infestations) | 7 | 8
Bronchitis (Infections and infestations) | 6 | 8
Impetigo (Infections and infestations) | 10 | 4
Viral infection (Infections and infestations) | 9 | 5
Pyrexia (General disorders) | 10 | 8
Fever (General disorders) | 12 | 0 — predefined term in subject diary; diary to be completed only by subjects receiving booster vaccination for 7 consecutive days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other